CLINICAL TRIAL: NCT00266981
Title: A Randomized Controlled Trial Which Compare the Effectiveness of an APOS Kit With Short Waves Therapy for Treating Whiplash Associated Disorders
Brief Title: Treatment of Whiplash Associated Disorders by APOS Kit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aposgo-HMO-CTIL
Record Dates: First submitted 2005-12-19; First posted 2005-12-20 (Estimated); Last update posted 2005-12-20 (Estimated); Status verified 2005-12

CONDITIONS: Whiplash Associated Disorders; Cervical Pain
MeSH Terms: conditions — Neck Pain

INTERVENTIONS:
Device: APOS - exercise component

SUMMARY:
The purpose of this study is to compare two techniques for treating patients with Whiplash Associated Disorders, in relation to: disability, balance, cervical pain and cervical range of motion.

The hypothesis: The APOS kit treatment is more effective than the short wave therapy.

ELIGIBILITY:
Inclusion Criteria:Cervical pain, Motor vehicle accident a week prior to cervical pain, age above 16, ability to walk independently, signed inform consent, insured in "Clalit health services" Exclusion Criteria: Inability to walk independently, age 16 or less, not signed an inform consent, WAD grade 4, past treatment for WAD, pregnancy, pacemaker, cancer.

-

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2006-03; Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
neck disability score
neck pain score
balance score
cervical range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Milka Donchin, MD, MPH, Principal Investigator — School of Public Health, Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel